CLINICAL TRIAL: NCT06661460
Title: Development and Preliminary Evaluation of a New Internet-Delivered Cognitive Behavioral Intervention for Youths With Anxiety Disorders
Brief Title: Internet-Delivered Cognitive Behavioral Intervention for Youths With Anxiety Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-04296-01
Record Dates: First submitted 2024-10-22; First posted 2024-10-28 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: ANXIETY DISORDERS (or Anxiety and Phobic Neuroses); Specific Phobia; Social Anxiety Disorder; Separation Anxiety Disorder; Generalized Anxiety Disorder; Panic Disorder; Agoraphobia
Keywords: Anxiety disorders; Children; Adolescents; Cognitive Behavioral Therapy; Remote delivery; Internet; Internet-delivered cognitive behavioral therapy
MeSH Terms: conditions — Anxiety Disorders; Phobic Disorders; Phobia, Specific; Phobia, Social; Anxiety, Separation; Generalized Anxiety Disorder; Panic Disorder; Agoraphobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-Delivered Cognitive-Behavioral Therapy (Experimental): Includes the intervention Internet-Delivered Cognitive-Behavioral Therapy.
  Interventions: Behavioral: Internet-Delivered Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Internet-Delivered Cognitive Behavioral Therapy — The intervention is a therapist-guided, internet-delivered cognitive behavioral therapy (ICBT) program primarily based on exposure therapy, involving the gradual confrontation of feared situations and/or stimuli. Treatment is accessed through a smartphone, tablet or laptop/desktop device. The 12-week intervention is available in two different versions depending on the participant's age: one for 8-12-year-olds and one for 13-17-year-olds. Each version consists of separate logins to 12 modules (chapters) for the child/adolescent and 12 modules for the caregivers. Both the child/adolescent and caregiver have individual contact with a trained therapist over the internet platform. The therapist provides feedback, responds to questions and sends reminders to complete the next module if required. Communication is carried out via text messages in the platform, via telephone (if deemed justified) and through a scheduled telephone or videoconference call approximately 4-5 weeks into treatment.

SUMMARY:
The goal of this study is to develop a new internet-delivered cognitive behavioral therapy (ICBT) intervention for youths with anxiety disorders based on the best current knowledge about effective cognitive behavioral therapy for the target group, refine the intervention in collaboration with patient and public representatives, and conduct a preliminary evaluation of the treatment effects in an open clinical trial.

The primary objective of the study is:

1. To evaluate the preliminary efficacy of a newly developed ICBT intervention for children and adolescents with anxiety disorders in reducing anxiety severity, as measured by the Pediatric Anxiety Rating Scale (PARS).

Secondary objectives of the study are:

1. To examine the preliminary efficacy (PARS) of the ICBT intervention at 3 months post-treatment.
2. To examine how youths with anxiety disorders, their caregivers, therapists, and healthcare leadership experience the ICBT intervention.
3. To examine factors (e.g., age, type of anxiety disorder, presence of depressive symptoms, experiences of ICBT) that predict treatment outcome.
4. To examine how the ICBT intervention can be improved (e.g., treatment content and technical delivery) for future use.

Participants will:

* Undergo ICBT treatment for anxiety disorders during 12 weeks
* Complete questionnaires at multiple time points throughout the study
* Participate in follow-ups post-treatment and 3 months post-treatment
* A selection of participants will also be invited to focus group interviews with the aim to generate ideas on how the intervention may be improved for future use

DETAILED DESCRIPTION:
A detailed description is available in the full study protocol. All full study protocol versions may be accessed at the Open Science Framework (https://osf.io/fdnga/).

ELIGIBILITY:
Inclusion Criteria:

1) 8 to <18 years of age.

* Confirmed by the child/caregiver and subsequently by the medical record system. 2) A principal DSM-5-TR anxiety disorder of specific phobia, separation anxiety disorder, social anxiety disorder, generalized anxiety disorder, panic disorder or agoraphobia.
* Confirmed by the Diagnostic Interview for Anxiety, Mood, and OCD and related Neuropsychiatric Disorders - Child and Adolescent Version (DIAMOND-KID).

  3) Child and caregiver able to read, write and communicate in Swedish.
* Confirmed by the child/caregiver. 4) An available caregiver who can support the child in treatment.
* Confirmed by the caregiver. 5) Access to a smartphone, tablet, or laptop/desktop device, and the internet.
* Confirmed by the child/caregiver.

Exclusion Criteria:

1) Principal DSM-5-TR anxiety disorder of specific phobia concerning the domain of blood-injection-injury (due to the ICBT program not including relevant information on applied-tension techniques to avoid fainting during exposure exercises).

* Confirmed by a blood-injection-injury phobia being classified as the principal anxiety disorder as assessed by the DIAMOND-KID.

  2) Established or suspected intellectual disability.
* Confirmed by the caregiver (through previous diagnosis) and/or by attending a special needs school for learning difficulties.

  3) Another mental disorder in more immediate need of management than an anxiety disorder (e.g., schizophrenia spectrum and other psychotic disorders, bipolar disorder, anorexia nervosa, substance use disorders).
* According to the DIAMOND-KID and/or other available sources. 4) Social/familial/educational difficulties in more immediate need of management than an anxiety disorder.
* Confirmed by the assessor through information from the child/caregiver and/or other available sources.

  5) Immediate risk to self or others that require urgent attention, such as acute suicidality.
* Confirmed by the assessor through information from the child/caregiver and other available sources.

  6) Previous CBT for an anxiety disorder, defined as five or more sessions with a certified CBT therapist within the 12 months prior to assessment.
* Confirmed by the child/caregiver or the medical record system. 7) Ongoing psychological treatment for an anxiety disorder.
* Confirmed by the child/caregiver or the medical record system. 8) Initiation or adjustment of any psychotropic medication for anxiety (i.e., selective serotonin reuptake inhibitors, tricyclic antidepressants, serotonin-norepinephrine reuptake inhibitor or antipsychotics) within 8 weeks prior to assessment.
* Confirmed by the child/caregiver or the medical record system. 9) Participation in user involvement sessions in the present study.
* Confirmed by the researcher.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Pediatric Anxiety Rating Scale (PARS) | Baseline; post-treatment (window of 12 to 18 weeks post-enrollment); 3-months post-treatment (window of 23 to 31 weeks post-enrollment).
  Used to assess anxiety severity. Clinician-rated. The scale yields a score of 0 to 35, with higher scores indicating more severe anxiety.

SECONDARY OUTCOMES:
Diagnostic Interview for Anxiety, Mood, and OCD and Related Neuropsychiatric Disorders - Child and Adolescent Version (DIAMOND-KID) | Baseline; post-treatment (window of 12 to 18 weeks post-enrollment); 3-months post-treatment (window of 23 to 31 weeks post-enrollment).
  Used to assess anxiety disorders and psychiatric comorbidity at baseline and anxiety disorders and major depression at follow-ups. Clinician-rated.
Clinical Global Impression Scale - Severity (CGI-S) | Baseline; post-treatment (window of 12 to 18 weeks post-enrollment); 3-months post-treatment (window of 23 to 31 weeks post-enrollment).
  Used to assess overall anxiety severity. Clinician-rated. Ratings are reported on a seven-graded scale from 1 ("Normal, not at all ill") to 7 ("Among the most extremely ill patients").
Clinical Global Impression Scale - Improvement (CGI-I) | Baseline; post-treatment (window of 12 to 18 weeks post-enrollment); 3-months post-treatment (window of 23 to 31 weeks post-enrollment).
  Used to assess level of improvement compared to admission. Clinician-rated. This single item scale ranges from 1 ("Very much improved") to 7 ("Very much worse").
Children's Global Assessment Scale (CGAS) | Baseline; post-treatment (window of 12 to 18 weeks post-enrollment); 3-months post-treatment (window of 23 to 31 weeks post-enrollment).
  Used to assess global impairment. Clinician-rated. The CGAS is a single item scale that ranges from 1 to 100, with a higher value indicating better functioning.
Therapist time | Consecutively throughout the 12 week treatment period.
  Therapist time: preparation time, support time in platform, support time via telephone, support time via videoconference, and documentation time. Reported in minutes per participant per week for each variable as well as combined.
Module completion | Consecutively throughout the 12 week treatment period.
  Completion of modules in the internet platform for each child/adolescent and each caregiver. Ranges from 0 to 12 modules. Reported separately for children, adolescents, caregivers of children, and caregivers of adolescents.
Number of participants with concomitant interventions | Post-treatment (window of 12 to 18 weeks post-enrollment); 3-months post-treatment (window of 23 to 31 weeks post-enrollment).
  Used to assess potential other treatments during the study period. Clinician-rated.
Revised Child Anxiety and Depression Scale - Child version (RCADS-C) | Baseline; post-treatment (window of 12 to 18 weeks post-enrollment); 3-months post-treatment (window of 23 to 31 weeks post-enrollment).
  Used to assess anxiety symptoms. Child/adolescent-reported. The RCADS version used in the present study is the 47-item version which ranges from 0 to 141 points, with higher scores indicating more severe internalizing symptoms.
Child Anxiety Life Interference Scale - Revised - Child version (CALIS-R-C) | Baseline; post-treatment (window of 12 to 18 weeks post-enrollment); 3-months post-treatment (window of 23 to 31 weeks post-enrollment).
  Used to assess life interference and impairment associated with childhood anxiety. The scale ranges from 0 to 36 points, with higher scores indicating higher interference and impairment. Child/adolescent-reported.
Patient Health Questionnaire-2 (PHQ-2) | Baseline; 3, 6, and 9 weeks into treatment; post-treatment (window of 12 to 18 weeks post-enrollment); 3-months post-treatment (window of 23 to 31 weeks post-enrollment).
  Used to assess mood and anhedonia symptoms. Child/adolescent-reported. Scores range from 0 to 6 points, with higher scores indicating more severe internalizing symptoms.
Generalized Anxiety Disorder-2 (GAD-2) | Baseline; 3, 6, and 9 weeks into treatment; post-treatment (window of 12 to 18 weeks post-enrollment); 3-months post-treatment (window of 23 to 31 weeks post-enrollment).
  Used to assess anxiety symptoms. Child/adolescent-reported. Scores range from 0 to 6 points, with higher scores indicating more severe anxiety.
Well-being | Baseline; 3, 6, and 9 weeks into treatment; post-treatment (window of 12 to 18 weeks post-enrollment); 3-months post-treatment (window of 23 to 31 weeks post-enrollment).
  Used to assess well-being, operationalized as satisfaction with life, overall happiness, and how much the person would change about their life if they could. Child/adolescent-reported. Scores range from 3 to 33 points, with higher scores indicating higher well-being.
Mood and Feelings Questionnaire (MFQ) - Suicidality item | Baseline; 3, 6, and 9 weeks into treatment; post-treatment (window of 12 to 18 weeks post-enrollment); 3-months post-treatment (window of 23 to 31 weeks post-enrollment).
  Single item taken from the Mood and Feelings Questionnaire (MFQ) used to assess suicidal ideation. Child/adolescent-reported. Scores range from 0 to 3 points, with higher scores indicating higher suicidal ideation.
Experiences of CBT - Child version | Baseline; 3, 6, and 9 weeks into treatment; post-treatment (window of 12 to 18 weeks post-enrollment).
  Used to assess experiences of receiving CBT. Child/adolescent-reported. The scale consists of 7 items (baseline), 12 items (3, 6, and 9 weeks into treatment; post-treatment). The baseline version consists of two separate scores ranging from 5 to 50 points (higher scores indicate a better treatment experience) and from 2 to 20 points (higher scores indicate a higher level of distress and interference). The mid- and post-treatment versions consist of three separate scores ranging from 9 to 90 points (higher scores indicate a better treatment experience), from 2 to 20 points (higher scores indicate a higher level of distress and interference), and from 1 to 6 points (higher scores indicate more time spent on treatment).
Working alliance - Child version | 3, 6, and 9 weeks into treatment.
  Used to assess the participant's perceived working alliance with their therapist. Child/adolescent-reported. The scale ranges from 0 to 36 points, with higher scores indicating better working alliance.
Adverse events questionnaire - Child version (AEQ-C) | 3, 6, and 9 weeks into treatment; post-treatment (window of 12 to 18 weeks post-enrollment).
  Used to assess adverse events/effects. Child/adolescent-reported. The scale consists of 22 yes/no items (score range 0-22 points) with higher scores indicating more present adverse events. For each adverse event that is present, there is also a rating of whether the adverse event is thought to be related to the provided treatment (yes or no).
Client Satisfaction Questionnaire - Child version (CSQ-8-C) | Post-treatment (window of 12 to 18 weeks post-enrollment).
  Used to assess treatment satisfaction. Child/adolescent-reported. The scale ranges from 9 to 36 points, with higher scores indicating greater satisfaction.
Need for treatment - Child version | Baseline; post-treatment (window of 12 to 18 weeks post-enrollment); 3-months post-treatment (window of 23 to 31 weeks post-enrollment).
  Used to assess the need of treatment for anxiety symptoms. Child/adolescent-reported. This single item scale ranges from 0 to 5 points, with higher scores indicating a higher need for treatment.
Revised Child Anxiety and Depression Scale - Parent version (RCADS-P) | Baseline; post-treatment (window of 12 to 18 weeks post-enrollment); 3-months post-treatment (window of 23 to 31 weeks post-enrollment).
  Used to assess anxiety symptoms. Caregiver-reported. The RCADS version used in the present study is the 47-item version which ranges from 0 to 141 points, with higher scores indicating more severe internalizing symptoms.
Child Anxiety Life Interference Scale - Revised - Parent version (CALIS-R-P) | Baseline; post-treatment (window of 12 to 18 weeks post-enrollment); 3-months post-treatment (window of 23 to 31 weeks post-enrollment).
  Used to assess life interference and impairment associated with childhood anxiety. Caregiver-reported. The scale ranges from 0 to 36 points, with higher scores indicating higher interference and impairment.
Experiences of CBT - Parent version | Baseline; 3, 6, and 9 weeks into treatment; post-treatment (window of 12 to 18 weeks post-enrollment).
  Used to assess experiences of receiving CBT. Child/adolescent-reported. The scale consists of 7 items (baseline), 12 items (3, 6, and 9 weeks into treatment; post-treatment). The baseline version consists of two separate scores ranging from 5 to 50 points (higher scores indicate a better treatment experience) and from 2 to 20 points (higher scores indicate a higher level of distress and interference). The mid- and post-treatment versions consist of three separate scores ranging from 9 to 90 points (higher scores indicate a better treatment experience), from 2 to 20 points (higher scores indicate a higher level of distress and interference), and from 1 to 6 points (higher scores indicate more time spent on treatment).
Working alliance - Parent version | 3, 6, and 9 weeks into treatment.
  Used to assess the caregiver's perceived working alliance with their therapist. Caregiver-reported. The scale ranges from 0 to 36 points, with higher scores indicating better working alliance.
Adverse events questionnaire - Parent version (AEQ-P) | 3, 6, and 9 weeks into treatment; post-treatment (window of 12 to 18 weeks post-enrollment).
  Used to assess adverse events/effects. Parent-reported. The scale consists of 22 yes/no items (score range 0-22 points) with higher scores indicating more present adverse events. For each adverse event that is present, there is also a rating of whether the adverse event is thought to be related to the provided treatment (yes or no).
Client Satisfaction Questionnaire - Parent version (CSQ-8-P) | Post-treatment (window of 12 to 18 weeks post-enrollment).
  Used to assess treatment satisfaction. Caregiver-reported. The scale ranges from 9 to 36 points, with higher scores indicating greater satisfaction.
Need for treatment - Parent version | Baseline; post-treatment (window of 12 to 18 weeks post-enrollment); 3-months post-treatment (window of 23 to 31 weeks post-enrollment).
  Used to assess the need of treatment for anxiety symptoms. Caregiver-reported. This single item scale ranges from 0 to 5 points, with higher scores indicating a higher need for treatment.
Avoidance and Fusion Questionnaire for Youth (AFQ-Y8) | Baseline.
  Used to assess psychological inflexibility. Child/adolescent-reported. The scale ranges from 0 to 32 points, with higher scores indicating greater psychological inflexibility.
The Cognitive-attentional Syndrome Questionnaire (CAS-1) | Baseline.
  Used to assess dysfunctional metacognitive beliefs. Child/adolescent-reported. The questionnaire consists of four domains. Each item of the three first domains is scored on a 0-8 point scale. Each item of the fourth domain is score on 0-100 scale. Higher scores indicates more dysfunctional metacognitive beliefs.
Swanson, Nolan, and Pelham Rating Scale (SNAP-IV) | Baseline.
  Used to assess attention difficulties, hyperactivity, impulsivity, and oppositional symptoms. Caregiver-reported. Each item is scored from 0 to 3 points. The item scores are then summarized in domains: inattention (items 1-9), hyperactivity-impulsivity (items 11-19) and oppositional (items 21-28). Items 10, 20 and 29 are not included in any of the domains. Higher scores indicate greater attention difficulties, hyperactivity, impulsivity, and oppositional symptoms.
Core autism traits - Child version | Baseline.
  Used to assess core autism traits. Child/adolescent-reported. The scale ranges from 0 to 36 points, with higher scores indicating greater autism traits.
Core autism traits - Parent version | Baseline.
  Used to assess core autism traits. Caregiver-reported. The scale ranges from 0 to 36 points, with higher scores indicating greater autism traits.
Focus groups | From week 12 and onwards (no specified end date in the study protocol).
  Qualitative data will be gathered through focus group interviews with the aim of generating novel ideas on how to enhance the ICBT intervention to better suit its target group. Four different types of focus groups will be compiled from the open clinical trial participants: children aged 8-12 years, b) caregivers of these children; c) adolescents aged 13-17 years; and d) caregivers of these adolescents.

CONTACTS AND LOCATIONS:
Overall Officials: Per Andrén, PhD, Principal Investigator — Department of Clinical Sciences, Lund, Lund University
Locations (1):
- Barn- och ungdomshälsan, Länssjukhuset, Kalmar, Region Kalmar Län, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
The data are pseudonymized according to national (Swedish) and European Union legislation and cannot be anonymized and published in an open repository. Participants in the study consent for their data to be shared with other international researchers for research purposes. The data can be made available upon reasonable request on a case-by-case basis according to the current legislation and ethical permits.

REFERENCES:
- See also: All full study protocol versions are published at the Open Science Framework (OSF). — https://osf.io/fdnga/